CLINICAL TRIAL: NCT01553032
Title: Skin Changes in Head and Neck Cancer During Immuno-(Chemo-) And Radiotherapy With Erbitux®
Brief Title: Skin Changes in Head and Neck Cancer During Immuno-(Chemo-) And Radiotherapy With Erbitux® (HICARE)
Acronym: HICARE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Heidelberg Medical Center (Other)
Collaborators: iOMEDICO AG (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Juergen Debus, Prof. Dr. Dr., University of Heidelberg Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UniHD-2010-11-40-1001; 2010-019748-38 (EudraCT Number)
Record Dates: First submitted 2011-05-31; First posted 2012-03-13 (Estimated); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Head and Neck Cancer
Keywords: Immuno-(Chemo-)and Radiotherapy; Erbitux®; Skin changes in Head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cetuximab; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erbitux® (Active Comparator)
  Interventions: Drug: Erbitux®
- Fractionated Radiotherapy (Active Comparator)
  Interventions: Radiation: Fractionated Radiotherapy

INTERVENTIONS:
Drug: Erbitux® — 400mg/m2 initial dose, followed by weekly doses of 250mg/m2 Treatment duration: 7-8 weeks
  Arms: Erbitux®
Radiation: Fractionated Radiotherapy — 30-35 fractions of radiotherapy (6-7 weeks)
  Other Names: 3D-conventional or IMRT
  Arms: Fractionated Radiotherapy

SUMMARY:
This is a national multicenter phase IV study to assess acute radiation dermatitis of combined radioimmuno(chemo)therapy with Cetuximab in patients with locally advanced, non-metastatic squamous cell carcinoma of the head and neck (LASCCHN).

DETAILED DESCRIPTION:
With the aim of optimizing combined treatment strategies in terms of efficacy as well as manageable side effects, the implementation of Cetuximab an EGFR targeting antibody demonstrated successfully a significant increase in survival times, although exhibiting an expected increase in skin toxicities (1,2). This Phase IV trial will explore this prominent side effect, which is due to a synergistic effect of radiodermatitis and acneiform rash, in great detail. In addition, feasibility aspects of the complex treatment schedule in common routine and with patients presenting an increased comorbidity rate compared to the study population studied in the pivotal Phase III trial will be observed.

Further, peripheral blood samples of patients that consent to participate in the molecular monitoring will be collected and their genetic, epigenetic- and transcriptional profiles correlated with clinical outcome parameters. The goal of this translational program is to identify and confirm novel peripheral blood based molecular predictors and surrogates of therapy response. Tissue samples and available medical evidence of patients that consent to participate in the assessment of the HPV status will be collected. The goal of this program is to correlate HPV status with clinical outcome parameters.

In addition, all patients will answer Quality of Life questionnaires including the EORTC QLQ-C30 questionnaire, the Head and Neck cancer specific module (3) and the Dermatology Life Quality Index (DLQI).

This prospective, open, multicenter phase IV study is designed to assess the rate of radiodermatitis in patients with LASCCHN treated with a combination of radiotherapy and the EGFR-targeted monoclonal antibody Cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, locally advanced (stage III, IVA or IVB) non-metastatic squamous-cell carcinoma of the oral cavity, oro- or hypopharynx and larynx
* ECOG Performance Status of 0-2
* ≥ 18 years of age
* Life expectancy of at least 6 months.
* Adequate bone marrow, liver and renal function (according to SmPC of Cetuximab) based on laboratory assessments raised within 7 days prior to start of study treatment.
* Signed and dated informed consent before the start of specific protocol procedures.
* Women of childbearing potential must have had a negative serum or urine beta-HCG pregnancy test within 7 days prior to the first administration of study treatment or must have a documented condition that prohibits pregnancy (e.g. post-menopausal; hysterectomy).
* Patients enrolled in this trial must be willing to use effective birth control measures during the course of the trial and the subsequent 2 months

Exclusion Criteria:

* Nasopharyngeal carcinoma
* Distant metastases
* Previous radiotherapy for carcinoma of the head and neck
* Participation in other clinical trial (according to the German Drug Law (Arzneimittelgesetz - AMG) within 30 days prior to start of study treatment
* Previous exposure to epidermal growth factor (EGFR) targeted therapy
* Known hypersensitive reaction to any of the components of study treatments
* Previous or concurrent cancer within 5 years prior to study entry that is distinct in primary site or histology except adequately treated basal cell carcinoma or preinvasive cervical carcinoma.
* Pregnant or breast-feeding patients
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results as judged by the investigator
* Any condition that is unstable or could jeopardise the safety of the patient and their compliance in the study as judged by the investigator
* Incapacity to consent or limited legal capacity to consent

Note: A combination of the applied radioimmunotherapy with a chemotherapy in terms of a Radioimmunochemotherapy (e.g. with Cisplatin or Carboplatin/5-Fluorouracil) is no exclusion criteria. Furthermore, a patient previously treated with an induction chemotherapy is allowed to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Rate of radiation dermatitis Grade 3/4 | 2 years after LPI
  Criteria for Adverse Events v4.0 (CTCAE) Grade 1: Mild Grade 2: Moderate Grade 3: Severe Grade 4: Life-theatening consequences Grade 5: Death

SECONDARY OUTCOMES:
Rate of radiation dermatitis Grade1/2 | 2 years after LPI
  Criteria for Adverse Events v4.0 (CTCAE) Grade 1: Mild Grade 2: Moderate Grade 3: Severe Grade 4: Life-theatening consequences Grade 5: Death
Rate of cetuximab-mediated acneiform rash Grade 1-4 | 2 years after LPI
  Criteria for Adverse Events v4.0 (CTCAE) Grade 1: Mild Grade 2: Moderate Grade 3: Severe Grade 4: Life-theatening consequences Grade 5: Death
Rate of cetuximab-mediated rhagades | 2 years after LPI
  Criteria for Adverse Events v4.0 (CTCAE) Grade 1: Mild Grade 2: Moderate Grade 3: Severe Grade 4: Life-theatening consequences Grade 5: Death
Rate of cetuximab-mediated nail changes | 2 years after LPI
  Criteria for Adverse Events v4.0 (CTCAE) Grade 1: Mild Grade 2: Moderate Grade 3: Severe Grade 4: Life-theatening consequences Grade 5: Death
ORR; LRC; PFS; OS | 2 years after LPI
  In %
Safety profile | 2 years after LPI
Median dose density of radiation | 2 years after LPI
Safety profile of applied radiation protocol | 2 years after LPI

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Debus, Prof. Dr. Dr, Principal Investigator — University Heidelberg, Klinik für Radioonkologie und Strahlentherapie, Im Neuenheimer Feld 400, 69120 Heidelberg
Locations (1):
- University of Heidelberg Medical Center, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Habl G, Potthoff K, Haefner MF, Abdollahi A, Hassel JC, Boller E, Indorf M, Debus J. Differentiation of irradiation and cetuximab induced skin reactions in patients with locally advanced head and neck cancer undergoing radioimmunotherapy: the HICARE protocol (head and neck cancer: immunochemo and radiotherapy with erbitux) - a multicenter phase IV trial. BMC Cancer. 2013 Jul 15;13:345. doi: 10.1186/1471-2407-13-345. PMID 23855804